CLINICAL TRIAL: NCT05024695
Title: A Prospective, Multicenter Masked Clinical Trial to Evaluate the Safety and Effectiveness of the MINIject CS627 Implant in Subjects With Open Angle Glaucoma
Brief Title: Evaluate the Safety and Effectiveness of iSTAR Medical's MINIject™ Implant for Lowering Intraocular Pressure (IOP) in Subjects With Primary Open-angle Glaucoma.
Acronym: STAR-V
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: iSTAR Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISM06 (STAR-V)
Record Dates: First submitted 2021-08-23; First posted 2021-08-27 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-06

CONDITIONS: Glaucoma
Keywords: glaucoma; MIGS; primary open angle glaucoma; suprachoroidal space; supraciliary space
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle; Choroidal Effusions

STUDY DESIGN:
Masking Description: Person(s) checking intraocular pressures are masked, except for day of surgery, throughout the duration of the trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Implant Group (Experimental)
  Interventions: Device: MINIject™ Implant

INTERVENTIONS:
Device: MINIject™ Implant — The MINIject™ SO627 is an integrated system for Minimally Invasive Glaucoma Surgery (MIGS) comprised of a glaucoma drainage implant, the MINIject™ SO627 and the SO Delivery System, designed to deliver the MINIject™ implant into the supraciliary space.

SUMMARY:
Evaluate the safety and effectiveness of iSTAR Medical's MINIject™ implant for lowering intraocular pressure (IOP) in subjects with primary open-angle glaucoma.

DETAILED DESCRIPTION:
This is a prospective, multicenter, masked clinical trial to evaluate the safety and effectiveness of iSTAR Medical's MINIject™ implant for lowering intraocular pressure (IOP) in subjects with primary open-angle glaucoma.

ELIGIBILITY:
Key Inclusion Criteria:

* Males and females, 46 years of age or older
* A diagnosis of primary open-angle glaucoma, who are candidates for medical therapy, laser treatment, or glaucoma-filtering surgery
* Pseudophakic with prior uncomplicated cataract surgery

Key Exclusion Criteria:

* Angle closure, congenital, or secondary glaucoma
* Diagnosed degenerative visual disorders
* Clinically significant intraocular inflammation or infection

Min Age: 46 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 975 (Estimated)
Dates: Start 2021-08-19 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure decrease | 24 months
  Proportion of subjects with ≥ 20% decrease (responders) from Baseline in unmedicated Diurnal IOP at Month 24.
Intraocular pressure decrease (outcome 2) | 24 months
  Change from baseline in mean unmedicated diurnal IOP at Month 24.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Glibert, Study Director — iSTAR Medical
Locations (37):
- United States (28):
  - Arizona Advanced Eye Research Institute, Glendale, Arizona
  - Vold Vision, Fayetteville, Arkansas
  - Beverly Hills Institute of Ophthalmology, Beverly Hills, California
  - Reeve Woods Eye Center, Chico, California
  - Sacramento Eye Consultants, A Medical Corporation, Sacramento, California
  - Grand Junction Eye Care, Grand Junction, Colorado
  - Eye Associates of Fort Myers, Fort Myers, Florida
  - Intermountain Eye Center, Eagle, Idaho
  - Illinois Eye Center, Peoria, Illinois
  - Virdi Eye Clinic, Rock Island, Illinois
  - Stiles Eyecare Excellene and Glaucoma Institute, Overland Park, Kansas
  - LA Eye and Laser, Alexandria, Louisiana
  - Minnesota Eye Consultants, Bloomington, Minnesota
  - Eye Consultants PC, Omaha, Nebraska
  - Center for Sight Las Vegas, Las Vegas, Nevada
  - NYU Langone Ophthalmology, New York, New York
  - Apex Eye Clinical Research, LLC, Mason, Ohio
  - Oklahoma Eye Surgeons, Oklahoma City, Oklahoma
  - Vanderbilt Eye Institute, Nashville, Tennessee
  - Glaucoma Associates of Texas, Dallas, Texas
  - El Paso Eye Surgeons, El Paso, Texas
  - Ophthalmology Associates, Fort Worth, Texas
  - Houston Eye Associates, Houston, Texas
  - Berkeley Eye Center, Houston, Texas
  - R and R Eye Research, San Antonio, Texas
  - The Eye Institute of Utah, Salt Lake City, Utah
  - Spokane Eye Clinical Research, Spokane, Washington
  - Eye Centers of Racine and Kenosha, Kenosha, Wisconsin
- Canada (3):
  - Prism Eye Institute, Oakville, Ontario
  - The Institute de l'Oeil des Laurentides, Boisbriand, Quebec
  - Clinique Opthalmologies Bellevue, Montreal
- Swiss Glaucoma Research Foundation Swiss Visio Montchoisi, Lausanne, Switzerland
- United Kingdom (5):
  - Queen Victoria Hospital NHS Foundation Trust, East Grinstead
  - Glaucoma Service Moorfields Eye Hospital, London
  - Imperial College Healthcare NHS Trust Western Eye Hospital, London
  - KCL Frost Eye Research Department St Thomas' Hospital, London
  - Research & Development Unit, Learning and Research Centre (LaRC), York Hospital, York

IPD SHARING:
Plan to Share IPD: No